CLINICAL TRIAL: NCT05262348
Title: A Prospective, Multi-center, Open-label, Pivotal Clinical Trial to Compare the Safety and Effectiveness of Adaptive Versus Conventional Stimulation in Advanced Levodopa-Responsive Parkinson's Disease Treated With Bilateral Deep Brain Stimulation
Brief Title: An Open-label Clinical Trial to Compare the Safety and Effectiveness of Adaptive Versus Conventional Deep Brain Stimulation
Acronym: ADVENT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study design has been revised and this protocol was never activated.
Sponsor: Newronika (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NWK_AlphaDBS_PIV_2022
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1a - conventional stimulation (Active Comparator): Stimulation will be delivered bilaterally to the STN or the GPi. The stimulation parameters will be based upon standard practice by the neurologist.
  Interventions: Device: conventional DBS delivered through AlphaDBS IPG System
- Phase 1b - adaptive stimulation (Experimental): Stimulation will be delivered bilaterally to the STN or the GPi, with the neurologist-set therapeutic window (which corresponds to the upper and lower limits for aDBS amplitude). The stimulation will be automatically adapted according to the personalized algorithm based on real time LFP analysis.
  Interventions: Device: adaptive DBS delivered through AlphaDBS IPG System

INTERVENTIONS:
Device: adaptive DBS delivered through AlphaDBS IPG System — The AlphaDBS IPG System delivers both conventional DBS and adaptive DBS. Adaptive DBS is a programming mode that provides stimulation in a closed-loop adaptive "real-time" fashion, using a biosignal recorded from the same macro-electrodes routinely implanted for DBS as an input variable.
  Other Names: aDBS
  Arms: Phase 1b - adaptive stimulation
Device: conventional DBS delivered through AlphaDBS IPG System — The AlphaDBS IPG System delivers both conventional DBS and adaptive DBS. Conventional DBS is programmed by DBS specialists.
  Other Names: cDBS
  Arms: Phase 1a - conventional stimulation

SUMMARY:
The clinical trial aims to evaluate the safety and effectiveness of bilateral subthalamic nucleus (STN) and Globus Pallidus internus (GPi) deep brain stimulation (DBS) with the AlphaDBS IPG System when programmed in adaptive versus conventional stimulating modes. It includes an initial open-label, crossover phase and a long term follow-up phase, during which the patient is free to switch between stimulating modes.

DETAILED DESCRIPTION:
This is an international multi-center (North America and Europe) clinical trial to evaluate the safety and effectiveness of bilateral STN and GPi DBS with the AlphaDBS IPG System when programmed in adaptive (aDBS) versus conventional (cDBS) stimulating modes, in patients with advanced levodopa-responsive Parkinson's disease (PD).

The protocol is comprised of:

Phase 1: Initial Treatment Period: Cross-Over Design

* Phase 1a: All patients will start the study in cDBS mode. After a 1-month post-surgical stabilization, the AlphaDBS IPG System will be turned ON in cDBS mode. Participants will complete a 1-month period of programming optimization (to fine tune medical therapies and stimulation parameters) followed by a 3-month period of cDBS.
* Phase 1b: At the end of the 3-month follow up in cDBS, participants will be switched to the aDBS mode. Participants will then complete a 1-month period of optimization (to fine tune medical therapies and stimulation parameters) followed by a 3-month period of aDBS.

Phase 2: Long-term follow-up: Naturalistic Follow-up Design Patients completing Phase 1 are eligible to enter long-term follow-up for up to an additional 28 months. During this time, patients are free to change the DBS mode as preferred (with a maximum switches set by the physician). Visits at 6-month follow-ups will collect safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥55 years old
2. Patient has been diagnosed with levodopa-responsive idiopathic Parkinson's disease for ≥5 years
3. The disease stage is II, III or IV according to the Hoehn and Yahr scale
4. Patient has history of improvement of Parkinson's symptoms as a direct result of administering levodopa
5. PD-related symptoms are not adequately controlled with medication, including motor complications of recent onset (>4 months duration)
6. Patient experiences persistent disabling PD-related symptoms or drug side effects (e.g., dyskinesia, motor fluctuations, or disabling "off periods") despite optimal medical therapy
7. Patient has been selected for bilateral STN or Gpi DBS, independently from this study, in accordance with local standard of care DBS screening
8. Patient has been selected to receive Medtronic leads model 3389 or 37086, independently from this study, in accordance with local standard of care DBS screening
9. Patient has DBS circuit integrity assessed and confirmed by impedance testing, before IPG implantation
10. ≥6 hours per day (waking hours) with poor motor symptoms control (time "OFF" plus time "ON" with dyskinesia) despite optimal medical therapy, as assessed by the 3-day diary
11. Montreal Cognitive Assessment (MoCA) >26 in MedON condition
12. Beck Depression Inventory II (BDI-II) score <17 in MedON condition
13. UPDRS-III improvement by ≥33% following intake of anti-parkinsonian medications
14. Patient is able to understand the study requirements and the treatment procedures and has provided written informed consent to participate
15. Patient is willing and capable of completing a 3-day diary and reaches a sufficient level of agreement (> 75%) with study personnel responses
16. Patient has a responsible caregiver who will help completing the 3-day diary, provide feedback on activities of daily living (ADL), and ensure the patient complies with visit schedule
17. Patient is willing to maintain a constant anti-PD medication treatment (best medical management) for at least one month prior to study enrollment
18. Patient is willing and able to attend all study-required visits, complete the study procedures and attend appropriate follow up visits

Exclusion Criteria:

1. Patient has contraindications for DBS surgery, including any intracranial abnormality (e.g., generalized atrophy, vascular malformation, hydrocephalus, hematoma, cavernous or venous angioma, tumor or metastases, midline shift, etc.) or metallic implant (e.g., aneurysm clip, cochlear implant, etc.)
2. Patient has a history of suicide attempt or current active suicidal ideation as determined by a positive response to Item 2-5 of suicide ideation sub-scale of the Columbia Suicide Severity Rating Scale (CSSR-S)
3. Patient has dementia, major depression, seizures, congestive heart failure, uncontrolled diabetes, dialysis, substance use disorders as described in DSM-V, or any other severe medical condition
4. Patient has any medical condition that could interfere with study procedures, confound the assessment of study endpoints, or prevent a proper data collection
5. Patient had confirmation of diagnosis of a terminal illness associated with survival <12 months
6. Patient needs repeated MRI scans
7. Patient requires diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT)
8. Patient carries an electrical or electromagnetic implant (e.g., cochlear prosthesis, pacemaker, neurostimulator, etc.)
9. Patient has, or plans to obtain, an implanted electrical stimulation medical device and/or an implanted medication pump (e.g., DUOPATM infusion pump) and/or is treated with a portable infusion pump
10. Patient is on anticoagulant therapy which cannot be paused for >5 days before IPG implant surgery
11. Patient with a history of cranial surgery including ablation procedure or any other previous neurosurgical procedure for the treatment of PD symptoms on either side of the brain
12. Patient is currently participating in another clinical study (excluding any sub-study of the present study)
13. Patient is a female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess Treatment-Emergent Adverse Events | 9 months
  To identify Treatment-Emergent Adverse Events (TEAEs) (including serious, device-related, stimulation-related, and/or procedure related TEAEs), discontinuations of aDBS and study discontinuation and physical or neurological findings as categorized by the Data and Safety Monitoring Board.
To compare change in Good on time (GOT) when the patient receives aDBS versus change in GOT when the patient receives cDBS. | 9 months
  The expected treatment effectiveness of AlphaDBS IPG System with aDBS mode (∆GOTaDBS = GOTaDBS@3-Months - GOT@Baseline) and with cDBS mode (∆GOTcDBS = GOTcDBS@3-Months - GOT@Baseline) will not differ more than two hours.

SECONDARY OUTCOMES:
Success rate, number of patients with at least 2 hours improvement in each treatment mode | 9 months
  Treatement success is defined as number of patients with >2 hours ∆GOTaDBS and ∆GOTcDBS
Patient fluctuations | 9 months and 36 months
  Number of ON/OFF transitions based on the 3-day diary
UPDRS III | 9 months and 36 months
  UPDRS III score, in MedOFF-StimON and MedON-StimON conditions
UdysRS | 9 months and 36 months
  Score of the Unified Dyskinesia Rating Scale (UdysRS) in MedOFF-StimON and MedON-StimON condition.
Percentage of time in which the system is used in aDBS mode | 28 months
  During the long term follow up, when the patient will be able to switch between programming modes, the patient preference will be assessed considering the percentage of time in which the system is used in aDBS.

IPD SHARING:
Plan to Share IPD: No